CLINICAL TRIAL: NCT05914883
Title: The NORwegian Atrial Fibrillation Self-SCREENing
Acronym: NORSCREEN
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: Sorlandet Hospital HF (Other Government); Haukeland University Hospital (Other); St. Olavs Hospital (Other); University Hospital of North Norway (Other)
Responsible Party: Principal Investigator, Sigrun Halvorsen, Professor, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 477781
Record Dates: First submitted 2023-06-08; First posted 2023-06-22 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to screening with continuous ECG screening for 3-7 days, or control/standard of care
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ECG screening (Experimental): ECG247 is used for continuous screening for 3-7 days
  Interventions: Diagnostic Test: Long-term continuous ECG monitoring
- No ECG screening (No Intervention): Standard of care

INTERVENTIONS:
Diagnostic Test: Long-term continuous ECG monitoring — Long-term continuous ECG monitoring with ECG247 Smart Heart Sensor
  Arms: ECG screening

SUMMARY:
Atrial fibrillation (AF) is common, increases the risk of mortality, stroke and heart failure, and portending significant burden to patients, societal health and health economy. One of three AF cases are undiagnosed. Several methods for detection of AF exist, but most of them have major limitations and are associated with resource-demanding diagnostic workup in the speciality health care services.

DETAILED DESCRIPTION:
This randomized clinical trial will evaluate whether self-screening for AF with the ECG247 patch monitor will reduce AF-related morbidity.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥65 years and minimum one other risk factor for stroke according to the CHA2DS2-VASc risk score: Age ≥75 years, Diabetes, Heart failure, Hypertension, Previous stroke/TIA and/or Vascular disease
* Informed consent for participation

Exclusion Criteria:

* History of AF (self-reported)
* Use of anticoagulation therapy
* Pacemaker/CRT device
* No smart phone

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 50000 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2029-12 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Stroke | 5 years
  percent per year

CONTACTS AND LOCATIONS:
Overall Officials: Sigrun Halvorsen, PhD, Study Chair — Oslo University Hospital
Locations (1):
- Oslo Unvirsity Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Boskovic M, Jortveit J, Haraldsen MB, Berge T, Engdahl J, Lochen ML, Schuster P, Sandberg EL, Grimsmo J, Atar D, Anfinsen OG, Pripp AH, Grenne BL, Halvorsen S. The NORwegian atrial fibrillation self-SCREENing (NORSCREEN) trial: rationale and design of a randomized controlled trial. Europace. 2024 Oct 3;26(10):euae228. doi: 10.1093/europace/euae228. PMID 39248170